CLINICAL TRIAL: NCT03320837
Title: Metabolomic Profile of Urine Samples From Neonates Fed Exclusively With Breast Milk as Compared With the Profile of Neonates Fed With an Infant Formula Enriched With Synbiotics
Brief Title: Metabolomic Profile of Urine Samples From Neonates Fed With Breast Milk and an Infant Formula Enriched With Synbiotics
Acronym: mtburnIFsynb
Status: Completed | Type: Observational
Sponsor: Rontis Hellas SA (Industry)
Collaborators: National and Kapodistrian University of Athens (Other); National Hellenic Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: metabolomicsurinesynbio3x36nmr
Record Dates: First submitted 2017-10-13; First posted 2017-10-25 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Infant Development
Keywords: metabolomics; microbiome; infant formula; synbiotics; urine samples; NMR analysis
MeSH Terms: interventions — Infant Formula; Milk, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Breastfeeding group: Infant are exclusively fed with breast milk
  Interventions: Other: Breast milk
- Mixed feeding group: Infants are fed with mixed nutrition with breast milk and Rontamil Complete 1®
  Interventions: Dietary Supplement: Infant formula; Other: Breast milk
- Infant formula group: Infant are fed exclusively with Rontamil Complete 1®
  Interventions: Dietary Supplement: Infant formula

INTERVENTIONS:
Dietary Supplement: Infant formula — Breast milk substitute containing synbiotics
  Groups: Infant formula group; Mixed feeding group
Other: Breast milk — Breast milk
  Groups: Breastfeeding group; Mixed feeding group

SUMMARY:
The aim of this trial is to verify - based on metabolomics and other anthropometric parameters - whether exclusive nutrition of infant formula enriched with synbiotics (probiotics B.lactis and prebiotics FOS), Long-Chain Polyunsaturated Fatty Acids (AA, DHA) and nucleotides, is comparable to breast milk and to mixed nutrition including breast milk together with the enriched infant formula.

DETAILED DESCRIPTION:
Normal full-term infants aged 0-28 days, from singlet pregnancy, born by vaginal delivery or by caesarian section, with Apgar score >7 in the 1st and 5th minute, not requiring resuscitation during delivery, and with a normal intrauterine growth, i.e. between 11th and 89th percentile (AGA- appropriate for gestational age). The mother's medical history should be free of any chronic diseases and allergies, while the gestation history should be free of any complications and of any pharmaceutical treatment administration prior to delivery.

Exclusion criteria: insufficient weight gain and/or semiology of possible allergy to cow milk, hospitalization in NICU (Neonatal Intensive Care Unit), treatment of breastfeeding mother having given birth recently or of the neonate with antibiotics after delivery.

Method: 36 Infants in exclusive breastfeeding, 36 infants feeding exclusively on infant formula with synbiotics and 36 infants following mixed nutrition with breast milk and infant formula with synbiotics, for a period of 3 months have been selected on randomized basis. For all these three groups, the anthropometric parameters should be measured (length, weight, head perimeter), since the first day of newborn's inclusion in the trial and at the age of 15 days, 2 and 3 months. Moreover, at the age of 15 days, 2 months, 3 months and on the infant's inclusion day in the trial, newborns-infants urine sample should be collected by the attending doctor using a ball of cotton inserted into the disposable diaper and with the aid of an aspiration syringe the urine sample (2-3 ml) will be transferred to a sterile vial and finally stored at -80 °C. Then frozen urine samples will be sent in batches to a contracted diagnostic center in order to examine the metabolic profile of the three diets described above (exclusive breastfeeding, infant formula with synbiotics and mixed nutrition with breast milk and infant formula with synbiotics), with the help of NMR and selectively liquid chromatography /mass spectrometry (LC/MS). This urine collection gives reliable results and can be used in infants without causing any discomfort or side-effect.

ELIGIBILITY:
Inclusion Criteria:

* Normal full-term infants aged 0-28 days,
* From singlet pregnancy,
* Born by vaginal delivery or by caesarian section, with Apgar score >7 in the 1st and 5th minute,
* Not requiring resuscitation during delivery, and with a normal intrauterine growth, i.e. between 11th and 89th percentile (AGA- appropriate for gestational age).

Exclusion Criteria:

* Insufficient weight gain and/or semiology of possible allergy to cow milk,
* Hospitalization in NICU (Neonatal Intensive Care Unit),
* Treatment of breastfeeding mother having given birth recently or of the neonate with antibiotics after delivery.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Metabolomic profile of urine samples | Newborn's age of 2 days
  Then frozen urine samples will be sent in batches to a contracted diagnostic center in order to examine the metabolic profile of the three diets described above (exclusive breastfeeding, Rontamil Complete 1® and mixed nutrition with breast milk and Rontamil Complete 1®), with the help of NMR and selectively liquid chromatography /mass spectrometry (LC/MS). This urine collection gives reliable results and can be used in infants without causing any discomfort or side-effect.
Metabolomic profile of urine samples | Newborn's age of 15 days
  Then frozen urine samples will be sent in batches to a contracted diagnostic center in order to examine the metabolic profile of the three diets described above (exclusive breastfeeding, Rontamil Complete 1® and mixed nutrition with breast milk and Rontamil Complete 1®), with the help of NMR and selectively liquid chromatography /mass spectrometry (LC/MS). This urine collection gives reliable results and can be used in infants without causing any discomfort or side-effect.
Metabolomic profile of urine samples | Newborn's age of 2 months
  Then frozen urine samples will be sent in batches to a contracted diagnostic center in order to examine the metabolic profile of the three diets described above (exclusive breastfeeding, Rontamil Complete 1® and mixed nutrition with breast milk and Rontamil Complete 1®), with the help of NMR and selectively liquid chromatography /mass spectrometry (LC/MS). This urine collection gives reliable results and can be used in infants without causing any discomfort or side-effect.
Metabolomic profile of urine samples | Newborn's age of 3 months
  Then frozen urine samples will be sent in batches to a contracted diagnostic center in order to examine the metabolic profile of the three diets described above (exclusive breastfeeding, Rontamil Complete 1® and mixed nutrition with breast milk and Rontamil Complete 1®), with the help of NMR and selectively liquid chromatography /mass spectrometry (LC/MS). This urine collection gives reliable results and can be used in infants without causing any discomfort or side-effect.

CONTACTS AND LOCATIONS:
Overall Officials: Nicoletta Iacovidou, PhD, Study Director — National and Kapodistrian University of Athens
Locations (1):
- Aretaieio Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided